CLINICAL TRIAL: NCT01240434
Title: Estudio Prospectivo Aleatorizado Simple Ciego Sobre la Incidencia de Hernias Incisionales en Los Orificios de Los trócares de Laparoscopia: Cierre aponeurótico Superficial Frente a cicatrización aponeurótica Sin Cierre
Brief Title: Randomized Prospective Trial on the Occurrence of Laparoscopic Trocar Site Hernias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Jesús Lago Oliver, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: cierrlaparosc001
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2006-03

CONDITIONS: The Aim of the Study is to Analyze the Incidence of Trocar Site Hernia (TSH); in Orifices Created by Trocars Measuring ≥10 mm in Diameter,; and to Determine Whether Closure of the External Fascial Layer Prevents; TSH and Potential Related Complications.
Keywords: trocar hernia closure laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fascia closure of the surgical trocars (Active Comparator): Arm in which all the surgical trocar orifices are closed by suturing the external fascia of the abdominal wall with a number 1 monofilament absorbable suture (Polydioxanone)
  Interventions: Procedure: Trocar site closure
- Trocar site without closure (No Intervention): All the orifices of the trocar site are left open, closing only the skin.
  Interventions: Procedure: Trocar site closure

INTERVENTIONS:
Procedure: Trocar site closure — The study has 2 arms: one in which all the ST orifices are closed by suturing the external fascia of the abdominal wall with a number 1 monofilament absorbable suture (Polydioxanone) (Group A), and another in which all the orifices of the ST are left open, closing only the skin (Group B).

SUMMARY:
The investigators perform a simple-blind randomized trial with two groups, one in which all the orifices are closed by suturing the external fascia of the abdominal wall (Group A), and another in which the orifices are left open, closing only the skin (Group B). Monitoring for trocar site hernia lasted 2 years from the intervention.

DETAILED DESCRIPTION:
This is a single-blind trial including all patients undergoing laparoscopic surgery performed by the same surgical team (5 surgeons) and for whom at least one "study trocar" (ST) id use. STs is define as blunt-tip trocars that are inserted blind, had a diameter of 11 mm or 12 mm, and are not enlarged during surgery. The investigators have not studied the Hasson trocar, as the defect it creates is surgeon-dependent and not uniform.

The investigators exclude patients presenting factors that affect the scarring process, such as malnutrition (serum proteins <5 g/dl), advanced cancer, perioperative hemodynamic instability, or prolonged treatment with corticosteroids. Orifices that are enlarged for specimen extraction are also excluded, although other orifices in the same patient are included.

The investigators exclude the following patients: those who are converted to open surgery, those who underwent a second intervention with an open technique during the early postoperative period, or those who are lost to follow-up. Patients who hace not an ST after surgery (mostly patients with only one ST that have to be enlarged for specimen extraction) are excluded from the trial.

The investigators randomize patients using a random table from Excel® for Windows XP®.

The trocars that the investigators use are Endopath Xcel (Ethicon Endo-Surgery, Puerto Rico, USA), which are 11 mm and 12 mm in diameter.

The study has 2 arms: one in which all the ST orifices are closed by suturing the external fascia of the abdominal wall with a number 1 monofilament absorbable suture (Polydioxanone) (Group A), and another in which all the orifices of the ST are left open, closing only the skin (Group B).

This trial has been approved by the corresponding ethics committee. All the patients signe their informed consent to participate in the trial before randomization.

Follow-up involve 2 postoperative contacts for each patient, the first during the first year after the operation, and the second 2 years after the intervention. These contacts are made by phone, and the patient is asked about any lumps or discomfort in the scar area. A positive answer is followed by an appointment for a detailed examination and, if necessary an abdominal ultrasound scan.

Demographics, diagnosis, and surgical technique is analyzed for each patient, as is hospital stay, morbidity, and the number of trocars and STs used with their size and location.

For the topographic analysis, the investigators divide the abdomen in 7 areas according to the different fascial layers of the abdominal wall (Figure 1).

The statistical analysis is performed using SPSS 11.5 for Windows.

ELIGIBILITY:
Inclusion Criteria:

All the patients undergoing laparoscopic surgery performed by the same surgical team (5 surgeons) and for whom at least one "study trocar" (ST) is used. STs is defined as blunt-tip trocars that are inserted blind, had a diameter of 11 mm or 12 mm, and are not enlarged during surgery.

Exclusion Criteria:

Hasson trocar Patients presenting factors that affect the scarring process, such as malnutrition (serum proteins <5 g/dl), advanced cancer, perioperative hemodynamic instability, or prolonged treatment with corticosteroids. Orifices that are enlarged for specimen extraction are also excluded, although other orifices in the same patient are included.

Patients who are converted to open surgery. Patients who did not have an ST after surgery (mostly patients with only one ST that had to be enlarged for specimen extraction) were excluded from the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2006-03; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The incidence of trocar site hernia

SECONDARY OUTCOMES:
The incidence of wound infections
  The secondary outcome measure try to relation surgical wound infection with surgical wound closure of the fascia and the incidence of trocar site hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Lago J, Serralta D, Garcia A, Martin J, Sanz M, Perez MD, Turegano F. Randomized prospective trial on the occurrence of laparoscopic trocar site hernias. J Laparoendosc Adv Surg Tech A. 2011 Nov;21(9):775-9. doi: 10.1089/lap.2011.0262. PMID 22050610